CLINICAL TRIAL: NCT01675895
Title: Addition of Lidocaine to Levobupivacaine Reduces Intrathecal Block Duration: Randomized Controlled Trial
Brief Title: Addition of Lidocaine to Levobupivacaine Reduces Intrathecal Block Duration
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, DILEK YAZICIOGLU, Principal investigator, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DİLEKLEVOBUPİVACAİNE
Record Dates: First submitted 2012-08-24; First posted 2012-08-30 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2012-12

CONDITIONS: Benign Prostate Hyperplasia
Keywords: Hyperbaric Levobupivacaine; İntrathecal; Lidocaine; TUR-P
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Levobupivacaine; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group Levobupivacaine lidocaine (Experimental): Group Levobupivacaine lidocaine Spinal anesthesia with 1.5 ml hyperbaric levobupivacaine (6.75 mg) + 0.3 ml 2 % lidocaine
  Interventions: Drug: Levobupivacaine lidocaine spinal anesthesia
- Group Control (Active Comparator): Group Control levobupivacaine spinal anesthesia with levobupivacaine (6.75 mg) + saline
  Interventions: Drug: levobupivacaine Spinal anesthesia

INTERVENTIONS:
Drug: Levobupivacaine lidocaine spinal anesthesia — Spinal anesthesia
  Other Names: Chirocaine; Lidocaine
  Arms: Group Levobupivacaine lidocaine
Drug: levobupivacaine Spinal anesthesia — spinal anesthesia
  Other Names: Chirocaine
  Arms: Group Control

SUMMARY:
The main objective was to test the hypothesis that adding lidocaine to hyperbaric levobupivacaine could change the duration of levobupivacaine spinal block.

DETAILED DESCRIPTION:
A satisfactory spinal anaesthesia requires both a fast onset and proper duration at the same time. Transurethral resection of the prostate (TUR-P) is a surgery of medium duration. The addition of lidocaine to hyperbaric bupivacaine shortens the duration of bupivacaine spinal block and therefore provides more rapid recovery. This property of lidocaine is not verified with other local anesthetics. Levobupivacaine is a S-enantiomer of racemic bupivacaine and is a long acting local anesthetic.The aim of this prospective randomized controlled study was to investigate this effect of lidocaine, with a local anesthetic other than bupivacaine. It was hypothesized that the duration of the intrathecal block could change when performed with hyperbaric levobupivacaine mixed with low dose lidocaine and this technique could be consistent for the duration of TUR-P surgery. Participants will be followed on the day of surgery for primary and secondary outcome measures and 3 days postoperatively for complications (TNS).

ELIGIBILITY:
Inclusion Criteria:

* elective transurethral resection of the prostate (TUR-P)

Exclusion Criteria:

* patients with contraindications for spinal anesthesia,
* known sensitivity to the study drugs,
* emergency cases, and
* patients who refused spinal anaesthesia were excluded

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
The duration of the spinal block (S1 regression of the block) | participanta will be followed on the operation day
  the time between the intrathecal injection and sensorial block regression to S1 dermatome, measured in minutes

SECONDARY OUTCOMES:
postoperative care unit stay | participants will be followed on the operation day
  the time between the patient entered the PACU and left the PACU (when the sensorial block was regressed to S1 dermatome and the patient fulfilled an Aldrete score higher or equal to 9), measured in minutes

OTHER OUTCOMES:
maximum block level | participants will be followed on the operation day
  the dermatomal level that the sensorial block reached, determined with the pin prick test, expressed with dermatomes

CONTACTS AND LOCATIONS:
Overall Officials: Taylan Akkaya, MD, Study Director — Ankara Diskapi Yildirim Beyazit Teaching and Research Hospital, Turkey.
Locations (1):
- Ankara Diskapi Yildirim Beyazit Teaching and Research Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Lee SJ, Bai SJ, Lee JS, Kim WO, Shin YS, Lee KY. The duration of intrathecal bupivacaine mixed with lidocaine. Anesth Analg. 2008 Sep;107(3):824-7. doi: 10.1213/ane.0b013e3181806149. PMID 18713891